CLINICAL TRIAL: NCT03359746
Title: Grazoprevir/Elbasvir for Treatment of Hepatitis C Virus Genotype 4 Post Kidney Transplant
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC # 2171 009
Record Dates: First submitted 2017-10-11; First posted 2017-12-02 (Actual); Last update posted 2017-12-02 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): This is a prospective, interventional, case-control study at King Faisal Specialist Hospital & Research Centre in post-renal transplant patients who are receiving Grazoprevir/Elbasvir combination. Data will be compared with matched historical controls, which will be selected according to the following matching criteria: age, time from transplant to initiation of therapy. Only patients who completed at least 48 weeks of pegylated Interferon + Ribavirin therapy in the control group and 12 weeks of therapy on the case group will be enrolled. Any patient who received at least one dose of Grazoprevir/Elbasvir combination will be included in the safety analysis.
  Interventions: Drug: Grazoprevir/Elbasvir

INTERVENTIONS:
Drug: Grazoprevir/Elbasvir — Medication for treatment of patient
  Other Names: No other intervention

SUMMARY:
This is a prospective, interventional, case-control study at King Faisal Specialist Hospital & Research Centre in post-renal transplant patients who are receiving Grazoprevir/Elbasvir combination. Data will be compared with matched historical controls, which will be selected according to the following matching criteria: age, time from transplant to initiation of therapy. Only patients who completed at least 48 weeks of pegylated Interferon + Ribavirin therapy in the control group and 12 weeks of therapy on the case group will be enrolled. Any patient who received at least one dose of Grazoprevir/Elbasvir combination will be included in the safety analysis.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the subject must be:

* Male or female > 18 years on the day of consent signature.
* Post renal transplant with stable graft function divided into 2 groups according to Creatinine Clearance (CrCl <30 mL/min Or CrCl ≥30 mL/min).
* Positive HCV infection post renal transplant defined as: Positive HCV RNA with documented HCV Genotype 4 (including those with mixed infections with Genotype 4 & Genotype 1 or Genotype 4 & Genotype 6).
* Fibro scan (Liver Elastography) performed prior to the baseline with evidence of chronic HCV infection.
* Liver Cirrhosis subjects may be included but will be limited to those with compensated liver disease (Child Pugh-A)
* Patient understands the study procedures, alternative treatments available, risks involved with the study and voluntarily agree to participate by giving written informed consent.
* Reproductive potential patient agrees to avoid becoming pregnant or impregnating a partner until at least 6 months after the last dose of medication. Acceptable methods of contraception (IUD or contraceptive rod implanted into the skin may, or combination of two: diaphragm with spermicide (cannot be used in conjunction with cervical cap/spermicide); cervical cap with spermicide (women only), male condom or female condom (cannot be used together), oral contraceptive pills: estrogen/progestine or progestin-only pill, contraceptive skin patch, vaginal contraceptive ring, or subcutaneous contraceptive injection. Abstinence can be used as a sole method of contraception if it is consistently employed and considered acceptable by the patient and Institutional Review Board.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

* Is under the age of legal consent, is mentally or legally incapacitated, has significant emotional problems at the time of pre-study screening visit or expected during the conduct of the study or has a history of a clinically significant psychiatric disorder which, in the opinion of the investigator, would interfere with the study procedures.
* Is infected with HCV Genotypes 1,2,3,5 or 6 except those with Genotype 1 or 6 with mixed infection with Genotype 4.
* Is co-infected with Hepatitis B Virus or HIV.
* Has evidence of decompensated liver disease manifested by the presence of or history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy or other signs or symptoms of advanced liver disease (Child Pugh-B or Child Pugh-C based on a platelet count below 75000 or an albumin below 3 g/dL)
* Pregnant or nursing female or male patient with pregnant female partner.
* Contraindications for Grazoprevir/Elbasvir.
* Is currently participating or has participated in a study with an investigational compound within 30 days of signing informed consent and is not willing to refrain from participating in another such study during the course of this study.
* Has any condition or pre-study laboratory abnormality, ECG abnormality, or history of any illness, which, according to the opinion of the investigator, might confound the results of the study or pose additional risk in administering the study drugs to the subject.
* Patient has not signed informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-12-15 (Estimated); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants achieving sustained virologic response at 12 weeks after the end of all treatment (SVR12) | 12 weeks after end of all therapy
  SVR12 was defined as HCV RNA below the lower limit of quantification (<LLOQ) at 12 weeks after the end of all study therapy. The primary efficacy hypothesis for this study is that the percentage of participants with Hepatitis C Virus (HCV) Genotype 4 post renal transplant achieving SVR12 with Grazoprevir/Elbasvir combination

SECONDARY OUTCOMES:
Percentage of participants with change in circulating HCV RNA during treatment and after treatment discontinuation as compared to baseline. | 12 weeks during therapy
  Hepatitis C viral load refers to the amount of hepatitis C virus in a person's blood. The results of this test (known as a viral RNA test or HCV RNA test) are usually expressed as International Units/mL (IU/mL) or RNA copies/mL. The percentage of participants with change in circulating HCV RNA during treatment and after treatment discontinuation as compared to baseline will be reported.
Percentage of participants with a decrease, no change, or increase between baseline and post treatment week 12 in kidney function as measured by Estimated Glomerular Filtration Rate and Albumin Creatinine Ratio (ACR) | 12 weeks during therapy
  Any worsening of a preexisting condition related to kidney function that was associated with the use of Elbasvir/Grazoprevir. The Percentage of participants with a decrease, no change, or increase between baseline and post treatment week 12 in kidney function as measured by Estimated Glomerular Filtration Rate and Albumin Creatinine Ratio (ACR) will be reported.
Percentage of participants experiencing acute kidney transplant rejection compared to historical control. | 12 weeks during therapy
  Any worsening of a preexisting condition related to kidney transplant rejection that was associated with the use of Elbasvir/Grazoprevir. The percentage of participants experiencing acute kidney transplant rejection compared to historical control will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Abaalkhail, Md, Study Chair — King Faisal Specialist Hospital & Research Centre, Riyadh

IPD SHARING:
Plan to Share IPD: Undecided